CLINICAL TRIAL: NCT05703295
Title: Oncologic Safety of Sentinel Node Biopsy in Clinically Palpable Axillary Lymph Node in Breast Cancer Patients
Brief Title: Oncologic Safety of Sentinel Lymph Node Biopsy in Clinically Palpable Axillary Lymph Node in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ibraheem Mohamed, Resident, Assiut University
Other Study IDs: Sentinel lymph node biopsy
Record Dates: First submitted 2023-01-13; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Sentinel Lymph Node Biopsy
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biopsy — Sentinel lymph node biopsy

SUMMARY:
Evaluation patients with palpable lymph node with breast cancer by sentinel lymph node biopsy and how to affect on the management of breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in females and the 3rd leading cause of cancer mortality. One of the important aspects of breast cancer management is axillary staging and the status of axillary lymph nodes is an important prognosticator that affects adjuvant treatment decisions in patients with early breast carcinoma. Sentinel lymph node biopsy (SLNB), is considered to be the standard of care for node negative breast cancer, as it can save patients from the complications of axillary lymph node dissection (ALND). These complications include lymphedema, arm stiffness, and neuralgia, all of which significantly affect the patient's quality of life and raise healthcare costs. It also allows accurate axillary staging with minimal morbidity. Oncologic outcomes in terms of disease-free survival, overall survival, and locoregional recurrence rate were similar in the SLNB alone versus the ALND group in patients with clinically node-negative axilla. In doing the SLNB, a combination of radioactive technetium-99m and blue bye technique is preferred to increase the SLN identification rate than using one technique in isolation. The rationale for performing upfront SLNB as routine for patients being treated for breast cancer should be challenged, for this our study aiming for evaluation of the role of sentinel lymph node biopsy in management of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age more than 18 years.
2. fit for surgery.
3. Patients with no previous breast surgery. .

Exclusion Criteria:

1. patients less than 18 years.
2. patients unfit for surgery .
3. patients with advanced breast cancer.
4. Patients with previous breast surgery.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All patients admitted to Assuit university hospitals more than 18 years old which candidate to sentinel lymph node biopsy during the time of the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Oncologic safety of sentinel node biopsy in clinically palpable axillary lymph node in breast cancer patients | baseline
  Evaluation patients with palpable lymph node with breast cancer by sentinel lymph node biopsy and how to affect on the management of breast cancer.

REFERENCES:
- [Background] Dixon JM. Sentinel Lymph Node Biopsy in Breast Cancer Surgery. Ann Surg Oncol. 2016 Oct;23(11):3426-3428. doi: 10.1245/s10434-016-5434-6. Epub 2016 Jul 22. No abstract available. PMID 27448117
- [Background] Qiu SQ, Zhang GJ, Jansen L, de Vries J, Schroder CP, de Vries EGE, van Dam GM. Evolution in sentinel lymph node biopsy in breast cancer. Crit Rev Oncol Hematol. 2018 Mar;123:83-94. doi: 10.1016/j.critrevonc.2017.09.010. Epub 2017 Sep 20. PMID 29482783